CLINICAL TRIAL: NCT06947772
Title: Effectiveness of Skill Building Education on Arteriovenous Fistula Self-Care Behaviors and Quality of Life of Patients on Hemodialysis
Brief Title: Skill Building Education of Arteriovenous-Fistula Self-Care Behaviors and Quality of Life of Patients on Hemodialysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shifa Tameer-e-Millat University (Other)
Responsible Party: Principal Investigator, Bushra Sultan, Assistant Professor, Shifa Tameer-e-Millat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 057-25
Record Dates: First submitted 2025-03-29; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease; Hemodialysis; Hemodialysis Access Failure
Keywords: Slef-care behaviors; hemodialysis; quality of life; arteriovenous fistula; Kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula; Kidney Diseases | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The randomize control trial (RCT) parallel design with the allocation ratio 1:1 will be employed to assess the effectiveness of a skill-building educational intervention on the self-care behaviors and quality of life of AVF in hemodialysis patients
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data analyst will assist with permuted block randomization procedure will be used to separate random scheme in both setting (A) and (B). The sealed envelopes will be prepared by data analyst, shuffled, numbered serial, and placed in a locked drawer in both units (A and B), and only research assistant can access it. After consenting and completing baseline assessment, the research assistant will open a sealed envelope to reveal the patient's group assignment. The patient will then be assigned to specific group accordingly. Research assistant will ensure that intervention and control groups' patients will have dialysis in separate rooms or wards to prevent contamination in intervention. The sealed envelop will be coded with numbers the research assistant will not know what these numbers mean.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Active Comparator): Skill building educational intervention will be implemented into two session. First is theoretical and other is practical. In theoretical session patients will be teach about the AVF self-care behavior. In practical session patient will be teach about how to monitor their AVF. Monitoring of AVF include the assessment of AVF. Assessment have three steps. Inspection, palpation and auscultation.
  Interventions: Behavioral: Skill building education
- usual care (No Intervention): Control group will receive usual care in the dialysis units.

INTERVENTIONS:
Behavioral: Skill building education — This intervention includes two session. theoretical and practical. In theroretical patient will be teahc about self-care of AVF and in oracticla session they learn how to monitor their AVF. monitoring have three part. inspection, palpation and auscultation
  Other Names: education
  Arms: Interventional

SUMMARY:
The purpose of this study is to assess the effectiveness of skill building educational interventions in improving the self-care behaviors and quality of life of AVF in hemodialysis patients. This study will address questions.

What is the effect of skill building education on the self-care behaviors of AVF care and quality of life in patients in patients undergoing hemodialysis treatment? A total 274 participants will be recruited from dialysis units of the study hospitals. Using random allocation 137 participants will be assigned to the control group and 137 to the intervention group. The intervention group will additionally receive a skill building education for improving their self-care behaviors and quality of life of AVF.

Researcher will implement skill building educational intervention in interventional group to enhance the self-care behaviors and quality of life. This intervention have two session, first is theoretical and another one is practical. The primary outcome of this study is AVF self-care behaviors and secondary outcome is quality of life related to AVF. This outcome will be assessed using the Self-care Behaviors Scale with Arteriovenous Fistula in Hemodialysis patients (ASBHD-AVF). The secondary outcome will be assessed using the Hemodialysis Access-related Quality of Life (HARQ) which is a self-administered tool develop by Nordyke.

The primary and secondary outcomes will be assessed at: baseline, after the completion of the intervention, and follow-up data will be collected at the second and sixth weeks after intervention is completed. Data will be analyzed using the Statistical Package of Social Science (SPSS) version 25. Descriptive statistics, means and standard deviations will be used for the continuous variables, while frequencies and percentages will be utilized for categorical demographic data (gender, educational level, hemodialysis frequency, items of self-care behavior scale, QOL). Normality of data will be check and applied test accordingly.

DETAILED DESCRIPTION:
Hemodialysis treatment requires vascular access. The AVF is a long-lasting and effective vascular access. Dysfunction of AVF leads to numerous complications such as infection, bleeding, stenosis, aneurysm, and thrombosis. Taking care of AVF, its cleanliness, maintenance, daily monitoring of AVF, and engaging in strengthening exercises and management can enhance the effectiveness of dialysis treatment.

The middle range theory of chronic illness is utilized for the development of this intervention that possesses three components: self-care maintenance, self-care monitoring, and self-care management. The most common AVF self-care maintenance instructions include refraining from applying pressure on the AVF, avoiding blood pressure monitoring and blood sampling from the AVF arm. The primary objective of self-care monitoring is to differentiate the normal anatomy and physiology from abnormal conditions or changes in the body. Recognizing the physical changes initiates the decision-making process regarding the necessary course of action. Routine monitoring of AVF blood flow can be accomplished by palpating the AVF site with the palm to detect the presence of a thrill. Additionally, the identification of bruit can be detected by auscultating/using a stethoscope. In self-care management, the patients can evaluate the treatment implementation. Patients who manage their self-care can improve their health status, and overall well-being, and enhance their quality of life.

The randomize control trial (RCT) parallel design with the allocation ratio 1:1 will be employed.

The control group will receive the routine care information at the hemodialysis units. The health care staff provides the usual routine care to patients during their regular dialysis procedures.

Intervention group will receive skills building education that include didactic and practical session Timing of the intervention will set based on the overall health status of patients. Each participant will receive individualized didactic instruction and personalized practical training before the dialysis procedure start. These two sessions will be delivered on separate days within the same week.

The didactic session. The purpose of this session is to educate patients on AVF self-care maintenance. Participants will explore the AVF concept, their perceptions of AVF, their current care practices, and the individual responsible for their AVF care at home. Next, patients will be educated on fistula, its functionality, its significance, and its impact on social, emotional and mental health. The session will conclude within a total duration of 25-30 minutes before the dialysis.

The practical session. The purpose of the practical session is to build skills that promote AVF self-care assessment and monitoring. The session will conclude within 20 to 25 minutes. In this session, participants will be shown how to assess and monitor AVF skill using a checklist. The assessment will be step-wise process starting with inspection, palpation and auscultation.

1. Inspection serves the purpose of identifying any situation that may compromise the AVF functioning.
2. Palpation serves the purpose of training the participants to identify the thrill of their fistula.
3. Auscultation serves the purpose of training the participants to listen the bruits sounds with a stethoscope. At the end of this session, participants will have a return demonstration of skill. Patients will be instructed to follow this assessment daily utilizing the provided checklist. The checklist will be provided to the patients in the Urdu language.

Follow-up. There will be two follow-up assessments: the 2nd, and 6th week post-intervention. Throughout the intervention and follow-up periods. Patients will be advised to complete the checklist daily after assessing their AVF. Daily assessment of the AVF using the checklist will serve to reinforce their behaviors. PI will conduct pilot testing of the intervention on 10% of the sample.

Participants will initially be recruited using consecutive sampling techniques. The sample size was calculated by using G* power. The parameters used for sample size calculation were: alpha= 0.05, β=0.15; power 1- β=0.85, with an allocation ratio of 1:1 and effect size =0.4. After adjusting the anticipated 20% attrition rate, the final calculated sample size will be 274 participants, with 137 in each group.

Consented patients will be randomized into a control group and experimental group through permuted block randomization by using the sealed envelopes. After consenting and completing baseline assessment, the research assistant will open a sealed envelope to reveal the patient's group assignment. The patient will then be assigned to specific group accordingly. Blinding will be implemented at two levels. First, baseline data will be collected before randomization to prevent bias in data collection and maintain patient blinding regarding their group assignment. Second, the PI will not be involved in the data collection process to ensure objectivity. A research assistant will be responsible for data collection process and an independent data analyst will perform the data analysis to further minimize potential biases.

Information will be collected on demographic sheet, on Charlton's Comorbidity Index, Self-care Behaviors Scale with Arteriovenous Fistula in Hemodialysis patients (ASBHD-AVF) and hemodialysis Access-related Quality of Life (HARQ) questionnaire.

The primary outcome of this study is AVF self-care behaviors. The ASBHD-AVF is a 16 items self- assessment scale developed by Sousa et al to assess the self-care behaviors of AVF of hemodialysis patients. The scale consists of two subscales: 1) management of signs and symptoms (6 items) and 2) prevention from complications (10 items). Response options consist of a five-point Likert scale ranging from 1 (never develop the self-care) to 5 (always develop the self-care). The minimum score is 16 and a maximum score is 80. A higher score reflects a higher frequency of self-care behaviors. The overall reported reliability of this tool is 0.72 and CVI is 1. Permission to use the tool was obtained from author.

The secondary outcome of this study is Quality of Life related to AVF. This outcome will be assessed using the Hemodialysis Access-related Quality of Life (HARQ) which is a self-administered tool develop by Nordyke. This tool includes six domains and specific scales are used to assess various domains that impact a patient's quality of life.

The ASBHD-AVF and the HARQ tools will be translated into Urdu and validated to ensure they are appropriately adapted to the local context according to the Sousa & Rojjanasrirat, guideline. Moreover, the tools will be pilot-tested on 10% of the population of the same setting and Cronbach alpha will be calculated.

The primary and secondary outcomes will be assessed at: baseline, after the completion of the intervention, and follow-up data will be collected at the second and sixth weeks after intervention is completed. Data will be analyzed using the Statistical Package of Social Science (SPSS) version 25. Descriptive statistics, means and standard deviations will be used for the continuous variables, (age, income, dialysis duration, AVF Duration) while frequencies and percentages will be utilized for categorical demographic data (gender, educational level, hemodialysis frequency, items of self-care behavior scale, QOL). The normality of the data will be checked and appropriate test will be applied accordingly.

Approval to conduct the study is obtained from the institutional review board (IRB) and the Ethical Committee of the institution (Shifa International Hospital). Furthermore, permission to collect patient data is obtained from the head of hemodialysis units. Permission for using the tools already have been taken from the authors. The participants' autonomy will be ensured by using informed consent. No known risks are involved in this research, and the benefits of the study will be explained. However, patients may feel overwhelmed during the data collection process. Data collection process will be scheduled and divided into two slots according to participant's ease. Patients will be allowed to ask any questions related to the study. A serial code instead of the participant's name will be assigned to participants' data sheets. Participants' identity will be kept confidential.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

The study will include patients:

1. diagnosed with end-stage renal disease on hemodialysis through an arteriovenous fistula
2. aged 18 years or above.
3. who can read and understand the Urdu language.

Exclusion Criteria:

Exclusion Criteria

The study will exclude patients:

1. having any physical or mental disabilities that can interfere with their capacity to perform daily life activities.
2. with any visual and hearing impairment. -

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of Self-Care Behaviors with AVF in Hemodialysis Patients (ASBHD-AVF) | 4 months
  Primary outcome of this study will be the assessment of self-care behaviors related to AVF in hemodialysis patients. The ASBHD-AVF is a 16 itme self-assessment scale develop by Sousa et al (2015) to assess self-care behaviors of AVF of hemodialysis patients. This scale consists of two sub scale: 1) Management of sign and symptom and 2) Prevention from complication. Response option consists of five point Likert scale ranging from 1(nevern develop the self-care)-5 (always develop the self-care). The minimum scores is 16 and maximum is 80.A higher scores reflect higher frequency of self-care behaviors. Permission of this tool is taken. The overall reported reliability is 0.72 and CVI is1.

SECONDARY OUTCOMES:
Hemodialysis Access-Related Quality of Life (HARQ) | 4 months
  The secondary outcome will be the assessment of AVF quality of life by using the Hemodialysis Access Related Quality of Life (HARQ). This is a self-administered tool develop by (Nordyke,2020). This tool include six domains and specific scales are used to assess various domains that impact a patient's quality of life: symptoms domain, emotional domain, physical functioning domain, social and role functioning domain, sleep domain, and care related burden domain. Permission of this tool is obtained from author.

CONTACTS AND LOCATIONS:
Overall Officials: Bushra Sultan, PhD, Principal Investigator — Shifa College of Nursing (STMU)
Locations (1):
- Shifa College of Nursing, Islamabad, Pakistan

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-04-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT06947772/Prot_SAP_ICF_000.pdf